CLINICAL TRIAL: NCT03861650
Title: The Effect of Bone Marrow Aspirate Concentrate on Bone Regenerate During Rapid Mandibular Distraction Osteogensis
Brief Title: Evaluation of Effect of Bone Marrow Aspirate Concentrate on Distracted Mandibular Bone Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasser Mohamed Nabil Ahmed Khirat El Hadidi (Other)
Responsible Party: Sponsor-Investigator, Yasser Mohamed Nabil Ahmed Khirat El Hadidi, Assistant Lecturer, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 392
Record Dates: First submitted 2019-02-27; First posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Hemifacial Microsomia; Distraction of Bone
Keywords: bone marrow aspirate concentrate; Hemifacial Microsomia; Distraction osteogenesis
MeSH Terms: conditions — Goldenhar Syndrome; Diastasis, Bone | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Case-control trial
Who Masked: Participant, Care Provider
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bone Marrow Aspirate Concentrate (Experimental): Bone Marrow Aspirate Concentrate is prepared from bone marrow by aspiration by wide bore needle and then prepared by centrifugation to get rich mix of MSCs to improve healing
  Interventions: Other: Bone Marrow Aspirate Concentrate
- Saline (Sham Comparator): Sham or placebo drug in the control group
  Interventions: Other: Saline

INTERVENTIONS:
Other: Bone Marrow Aspirate Concentrate — A rich MSCs prepration made by centrifugation and concentration of aspirated bone marrow
  Arms: Bone Marrow Aspirate Concentrate
Other: Saline — Physiological saline is added in control group to act as placebo
  Arms: Saline

SUMMARY:
Maxillofacial Distraction Osteogenesis (DO) has a lot of draw backs; mostly related to long distraction and consolidation time. Rapid rate DO was proposed to decrease the distraction time to avoid consequences of long procedure. The idea of the current study is to provide mesenchymal stem cells (MSCs) in form of Bone Marrow Aspirate Concentrate (BMAC) during rapid distraction to fasten and shorten consolidation. Methods: This trial was conducted on patients requiring mandibular DO. Patients were divided in two groups; control group in which distraction took place at a rate of 1.5 mm /day without any enhancement and study group in which distraction took place at rate of 1.5 mm /day and the distracted bone was enhanced by BMAC

DETAILED DESCRIPTION:
Material and Methods:

A prospective case-control trial was conducted on patients requiring mandibular distraction osteogenesis to assess the effect of BMAC on distracted bone quality. Evaluation of newly formed bone quantity and quality was done using a CBCT which was done post distractor removal as a part of routine follow up ( in agreement with European guidelines for the exposure to ionizing radiation) and evaluation of the bone quality was assessed by two examiners to provide interexaminer-reliability.

In order to evaluate the effect of BMAC on bone maturation and possibility of early removal of the distractor; which was not feasible in the clinical study due to the ethical concerns. Mechanical three point bending was applied on distracted mandible after 30 days following distraction to evaluate bone healing and mechanical strength of distracted bone. In addition to histological and radiographic evaluation.

Patients and methods:

Patient grouping and anesthetic technique:

Prospective case-control trial was conducted on patients requiring mandibular distraction osteogenesis. The research was reviewed by the ethical committee of author faculty. Patients were randomly allocated into one of the two groups (To avoid bias, each patient had a number, and this number was picked by the examiners (similar to a deck of shuffled cards) to assign the patient to his/her specific group. Control group (6 patients): control group in which distraction took place at a rate of 1.5 mm /day till planned length was obtained and only saline was injected in defect; based on the assumption that it has no effect on bone healing. Study group in which distraction took place at rate of 1.5 mm /day till planned length was obtained. Distracted bone was enhanced by injection of Bone Marrow Aspirate Concentrate (BMAC).

Anesthesia was induced with IV propofol (Aspen, Ireland), 1.5-2 mg/kg, fentanyl (ADVANZ Pharma, United Kingdom) 1.3 μ/kg and succinyl choline (Aspen, Ireland) 1mg/kg to facilitate nasotracheal intubation using armored tube. Anesthesia was maintained with isoflurane (AbbVie Ltd, United Kingdom) in oxygen and atracurium (Accord-UK Ltd, United Kingdom) in a dose of 0.3-0.6 mg/kg.

BMAC preparation and harvesting:

BMAC was harvested using the Ficoll protocol. Bone marrow was collected the iliac crest using bone marrow trocar. Phosphate buffered saline (PBS) was added to the aspirated bone marrow in a 4:1 ratio. The diluted bone marrow was titrated over Ficoll 400 (BIOCOLL; Biochrom GmbH, Germany), and the solution was centrifuged at a rate of 2,000 rpm for 20 minutes. The buffy layer pellet, which is rich in BMMSCs, was collected using a pipette. The Aspirated BMAC rich with MSCs was added to tissue culture flasks for till day 10 consolidation in DMEM (Thermo Fisher Scientific, United States) and high streptomycin-penicillin concentrate 10,000 U/mL (Sigma-Aldrich, United States); to be stored at -80 0C till injection at day 10 consolidation .

Surgical procedure An intraoal incision was performed similar to bilateral sagittal split osteotomy in the last molar area area to expose the mandibular body. A piezotome was used with copious saline irrigation; to perform the corticotomy to avoid nerve injury. The osteotomy was completed using a chisel and a mallet.

The bi-directional distractor was fixed using four 2.0 extra oral pins. Trial activation and deactivation were performed in operation room to be sure of osteotomy completion before wound closure. A topical antibacterial mouth was used throughout the entire distraction and consolidation period to decrease the risk of infection Postoperative phase and distraction protocol A topical antibacterial mouth was used throughout the entire distraction and consolidation period to decrease the risk of infection. Amoxicillin 875 mg. /clavulanic acid 125 mg (Augmentin, GSK, United Kingdom) capsules twice daily for five days to decrease risk of infection. Ibuprofen 600 mg (Mylan Products Limited, United Kingdom) Tablets twice daily for three days to control pain.

Distraction phase was performed after 5 days of latency. The rate was 1.5 mm per day till the planned chin position was achieved. In the study group, after 10 days of distraction, the prepared BMAC ( the average number of cells was 3 million) were injected in the distraction gap using an 18-gauge needle on days 10 of the consolidation. The control group had no enhancement and was considered as a negative control. The study and control groups underwent 6 months of consolidation after then the distractor pins were removed and CBCT was performed to evaluate the distraction procedure. In addition to the CBCT evaluation of distraction results the distracted bone maturation was evaluated.

Methods of assessment Using the CBCT (iCAT, USA) DICOM files evaluation of bone density was performed (at a fixed exposure value 84 Kv, 4 mA and 12 Sec ) to evaluate bone quality post distraction. Evaluation was done at three points located between pins marks. The first evaluation was done in exact center and other two readings were done 2mm before and 2mm after the central reading in the CT and average was calculated. Two examiners did evaluation to avoid bias and inter examiner reliability was measured to assess accuracy of the measurements

ELIGIBILITY:
Inclusion Criteria:

1. Patients free from any disease affecting bone formation of both sexes was included in the study.
2. Patients younger than 25 years old.
3. Patients included in the study were post traumatic patients, hemifacial microsomia, Treacher Collins and post ankylotic mandibular deformity.
4. Distraction range was between 15-20 mm.

Exclusion Criteria:

1. The presence of uncontrolled systemic disease.
2. Previous radiotherapy on head and neck region.
3. Chemotherapy within the past 12-month period.
4. An active infection at the distraction site.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2015-12-30 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Assessment of effect of BMAC on rapidly distracted bone quality | 6 months
  radiographically the bone density was assessed using CBCT of the patients to evaluate the effect of BMAC on bone maturation in term of increased bone density measured in Hounsfield unit as the increase in bone density indicates better healing and more bone maturation and justify addition of BMAC

IPD SHARING:
Plan to Share IPD: Undecided